CLINICAL TRIAL: NCT00572884
Title: CCRC:Identification and Development of Biological Markers of Human Exposure to the Insecticide Permethrin
Brief Title: Metabolism of the Insecticide Permethrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Bruce D. Hammock, University of California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200311123-8; DAMD17-01-1-0769; P42ES004699 (NIH)
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Pharmacokinetics; Metabolism
Keywords: permethrin; pyrethroid; pharmacokinetics; metabolism; accelerator mass spectrometry; human exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: permethrin insecticide — 25 mg neat carbon-14 labelled permethrin applied dermally in isopropyl alcohol, once for 8 hours containing 1 microcurie of carbon-14

SUMMARY:
Military personnel are exposed to the insecticide permethrin when using the DOD Insect Repellent System. A urinary metabolite of permethrin that is in high abundance and is relatively stable may be an ideal biomarker of exposure to this pesticide. Monitoring such a biomarker can prevent over-exposure. The objectives are to identify the most abundant human urinary metabolite following dermal exposure; to utilize this information to develop rapid laboratory-based and field portable methods to monitor the degree of an individual's exposure to permethrin.

DETAILED DESCRIPTION:
Permethrin is applied to the forearm of the subject and remains for 8 hours. The exposed area is then washed with soap and water several times. 24 hour urine samples are collected at daily intervals for 192 hours. Blood and saliva samples are taken at pre-dose, 1, 3, 6, 9 12, 24, 48, 72, 96, 120, 144, 168 and 192 hours. Subjects must return to the clinic daily to drop off urine collections and have blood and saliva samples taken.

ELIGIBILITY:
Inclusion Criteria:

* self-report healthy adult men and premenopausal women

Exclusion Criteria:

* unusual alcohol, drug, cigarette use for last 3 years
* unusual exercise program for last 3 years
* under the care of a physician for a disease
* participated in any radioactive drug study
* pregnant
* lactating
* people who rely more on their arm due to illness or injury
* people with neurological or musculoskeletal diseases
* use of permethrin in the last 6 months
* people who apply pesticides as their primary occupation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2006-02; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Concentration of individual metabolites in urine | 192 hours

SECONDARY OUTCOMES:
total carbon-14 in serum | 192 hours
Total carbon-14 in saliva | 192 hours
Total carbon-14 in urine samples | 192 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Hammock, PhD, Principal Investigator — University of California, Davis
Locations (1):
- CTSC Research Center, Mather, California, United States